CLINICAL TRIAL: NCT01308125
Title: PREPARE PICSO A Study To Evaluate The Safety And Feasibility Of Pressure-controlled Intermittent Coronary Sinus Occlusion (PICSO) In Patients With Coronary Artery Disease Undergoing Native Vessel Intervention
Brief Title: Safety And Feasibility Study Of Pressure-controlled Intermittent Coronary Sinus Occlusion (PICSO) In Patients With Coronary Artery Disease Undergoing Native Vessel Intervention
Acronym: PICSO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Miracor Medical SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP 2009-03 PREPARE PICSO
Record Dates: First submitted 2011-02-03; First posted 2011-03-03 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Stable Angina
Keywords: Stable Angina; Coronary artery disease; PCI; Reperfusion; Myocardial Infarction; collateral flow pressure index; CFpI; pressure controlled intermittent coronary sinus occlusion; PICSO
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: PICSO — * Baseline (hemodynamic) measurement
  * Intra coronary
  * Blood sampling
  * LAD occlusion: for 3 min or until pain with and without PICSO
  * Break recovery: the patient can recover from pain for 3 min
  * CFIp: by a ComboWire advanced in the center lumen of an occlusion balloon.
  * PICSO: start automatically and continued for 10 min.
  * PCI/PICSO: concomitantly for the whole duration of the PCI intervention.
  * 24h Follow up: additional blood samples every 6 hours (4 times)
  * 30 days follow up.
  Other Names: PICSO Impulse System; PICSO Impulse Console; PICSO Impulse Catheter

SUMMARY:
Pressure intermittent coronary sinus occlusion (PICSO) in patients with coronary artery disease improves collateral flow index to higher than 30%. PICSO used in this patient population is safe, feasible and effective. Safety, feasibility and effectiveness will be tested by periprocedural and logistic data.

DETAILED DESCRIPTION:
1 Background Good collateral flow in case of obstructive coronary artery disease and acute myocardial has beneficial effects on morbidity and mortality. Pressure controlled Intermittent Coronary Sinus Occlusion (PICSO) carries a promise of improving myocardial flow, decreasing microvascular obstruction and decreasing the rate of peri-procedural and acute myocardial infarction without the increased risk of bleeding such as is encountered with gp2b3a inhibitors. This study is designed to evaluate the safety and feasibility of PICSO in patients with stable coronary artery disease and experimental short coronary artery occlusion.

2. Objective The purpose of the study is to determine whether PICSO is safe and feasible with a femoral approach, and in what amount of cases PICSO is effective to increase collateral flow index (CFI). In this study an adapted collateral flow pressure index (CFpI) will be used and is calculated as the ratio of the distal LAD pressure during LAD balloon occlusion (PLADoccl.) and the Aortic pressure (Pao). CFI>30% has been shown in several studies to be a significant predictor of inducible ischemia as measured by intracoronary ST-segment changes. The study is a non-randomized single centre trial using a Bayesian statistical model.

3. Specific This study is a study in 10 elective patients with coronary artery disease assessing the safety and feasibility of adjunctive PICSO treatment during PCI using a femoral vein approach.

Together with the preclinical experience using the Miracor technology, we therefore believe that the planned cohort of 10 patients is sufficient to corroborate earlier experiences on the safety of the procedure as well as present technology.

For the effectiveness, 10 sets of measurements before and after the procedure in each patient will provide insight into the clinical significance since each patient will serve as her or his control.

Study end-points

3.1 Primary endpoints

1. Duration from successful femoral vein cannulation until successful placement of PICSO Impulse catheter into the Coronary Sinus.
2. Relative increase in collateral flow pressure index (CFpI) during LAD occlusion with and without PICSO.

3.2 Secondary endpoints

1. Number of patients reaching collateral flow pressure index (CFpI) higher than 30% during PICSO.
2. Quantitative evaluation of pre-condition effect on relative increase of CFpI.
3. The change of ST segment as recorded at Intra coronary ECG measures during balloon inflation.

3.3 Primary safety endpoints

1. The patients are hemodynamic stable during PICSO.
2. Elevation of coronary sinus pressure
3. The 30 days MACE is comparable to other patients undergoing PCI.

   1. Stroke
   2. Bleeding
   3. Inflammation
   4. New onset of an acute coronary syndrome or newly documented heart failure, requiring therapy or hospitalization
   5. Pulmonary embolism
   6. Coronary sinus permanent occlusion
   7. Death
   8. Other Adverse Events
4. No reported Adverse Events caused by PICSO

ELIGIBILITY:
Inclusion Criteria:

* Subjects (men or women) at least 18 years of age and
* Coronary artery disease as assessed by angiography and
* Clinical indication for PCI and
* Able to understand content of and willing to provide written informed consent

Exclusion Criteria:

* Active and or treated malignancies within 12 months prior to Visit 1
* Anatomical complications (e.g. The system in not able to effectively occlude the coronary sinus)
* Presence of significant colleteral flow supplying the target vessel (Rentrop >1)
* Any significant systemic illness or medical condition that could lead to difficulty complying with the protocol; or any concurrent condition(s) which, in the investigator's opinion, would prohibit the subject from completing the study, or would not be in the best interest of the subject
* Bleeding or perforation during PCI, pericardial effusion and/or hematoma
* Cardiac arrest or arrhythmia requiring chest compressions or cardiopulmonary resuscitation
* Cardiogenic shock (Cardiac Index <1.8 L/min/meter-squared or as assessed by the investigator), pulmonary edema (Killip Class >2), or hemodynamic instability as assessed by the investigator at the time of cardiac catheterization
* Clinically significant renal disturbance (sMDRD calculated GFR≤30 mL/min/1,73m2)
* Coronary Sinus electrode in place
* Acute ST elevation myocardial infarction
* Previous Q-wave myocardial infarction in the target area
* History of acute myocardial infarction within 72h prior to screening
* Ejection fraction <20%
* History of stroke, any sequelae of a transient ischemic attack (TIA), reversible ischemic neurological defect (RIND) within 6 months prior to screening
* Left Bundle Branch Block
* Mitral regurgitation (MR) > grade I
* Mitral stenosis.
* Patient not currently in sinus rhythm
* Patients on cardiac resynchronization therapy (CRT) or scheduled for CRT implantation
* Patients with previous CABG or planned chronic total occlusion revascularization
* Pregnancy or active breast-feeding. Urine pregnancy tests will be performed on all women who are not post-menopausal for at least 1 year
* Registration in another interventional study
* Severe anemia at baseline (Hemoglobin <10 g/dl or <6.2 mmol/l)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
No reported Adverse Events caused by PICSO | 30 days

SECONDARY OUTCOMES:
The 30 days MACE is comparable to other patients undergoing PCI. | 30 days after intervention
  Number of patients of reported ADE described as:
  1. Stroke
  2. Bleeding
  3. Inflammation
  4. New onset of an acute coronary syndrome or newly documented heart failure, requiring therapy or hospitalization
  5. Pulmonary embolism
  6. Coronary sinus permanent occlusion
  7. Death
  8. Other Adverse Events
The patients are hemodynamic stable during PICSO. | 6 hours (during the whole intervention)
  The hemodynamic is constantly monitored during the whole intervention and will be qualified by:
  Arterial pressure, LAD pressure, LAD velocity, Coronary Sinus pressure, ECG
Relative increase in collateral flow pressure index (CFpI) during LAD occlusion with and without PICSO. | 6 hours (during the whole intervention)
  A ComboWire (VolcanoCorp, CA, USA) will be advanced in the center lumen of an occlusion balloon. This will allow performing the measurements below the experimental occlusion.
The change of ST segment as recorded at Intra coronary ECG measures during balloon inflation. | 6 hours (during the whole intervention)
  The presence or absence of ECG signs of myocardial ischemia during balloon occlusion will also be assessed on-line by means of the ST segment changes >0.1mV present on an intracoronary ECG lead obtained from the angioplasty guide wire placed distal to the stent (outside the OTW balloon) in the region on interest.
Number of patients reaching collateral flow pressure index (CFpI) higher than 30% during PICSO. | 6 hours (during the whole intervention)
  A ComboWire (VolcanoCorp, CA, USA) will be advanced in the center lumen of an occlusion balloon. This will allow performing the measurements below the experimental occlusion, see also above.
Quantitative evaluation of pre-condition effect on relative increase of CFpI. | 6 hours (during the whole intervention)
  A ComboWire (VolcanoCorp, CA, USA) will be advanced in the center lumen of an occlusion balloon. This will allow performing the measurements below the experimental occlusion. A comparision will be made between the LAD occlusion phase with or without PICSO.
Duration from successful femoral vein cannulation until successful placement of PICSO Impulse catheter into the Coronary Sinus. | 1 hours (at the begin of the intervention)
  For each case the time will be captured and the average time will be calculated from all enrolled cases.
Intermittent elevation of coronary sinus pressure | 6 hours (during the whole intervention)
  The coronary sinus pressure will be recorded during the whole intervention. The relative mean and max. increase during the PICSO-phase will be evaluated per Patient and over all cases.

CONTACTS AND LOCATIONS:
Overall Officials: Jan J. Piek, Prof, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center Amsterdam, Amsterdam, Netherlands